CLINICAL TRIAL: NCT03706846
Title: Study of Two Fasting Procedures Before Gastroscopy: 6 Hours Versus 2 Hours for Clear Fluids
Acronym: GASTROPREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P/2017/343
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; Upper digestive endoscopy; fasting; esophageal cancer; Superficial neoplastic lesions; Esophageal mucosa; Gastric mucosa
MeSH Terms: conditions — Fibrosis; Fasting; Esophageal Neoplasms | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting 2 hours (Other): Fasting 2 hours
  Interventions: Procedure: fasting
- Fasting 6 hours (Other): Fasting 6 hours
  Interventions: Procedure: fasting

INTERVENTIONS:
Procedure: fasting — fasting before gastrointestinal endoscopy

SUMMARY:
Upper gastrointestinal endoscopy is the key examination for screening for precancerous and cancerous lesions of the esophagus and stomach. This study aims to describe the quality of the visualization of the esophageal and gastric mucosa, the safety of use of two fasting procedures before gastroscopy and the feeling of patients. The population evaluated here concerns cirrhotic patients, at high risk of developing a precancerous lesion of the upper gastrointestinal tract.

The investigator carries out a prospective, monocentric (Besançon CHRU), interventional and randomized study according to two fasting procedures before gastroscopy: 6 hours (F6 group) versus 2 hours (F2 group) for clear fluids. The primary endpoint was to describe and compare the quality of visualization of the esophageal and gastric mucosa, graded from A (good quality) to C (poor quality) according to a score. developed by Elvas et al. (Endoscopy 2017).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Male or female
* Cirrhosis based on radiological, clinical, biological or histological criteria

Exclusion Criteria:

* Diabetes for more than 10 years;
* Under 18 years of age;
* History of inhalation
* Patients in whom the gastrointestinal anatomy has not been retained
* Subjects who were unlikely to cooperate with the study and / or in whom poor cooperation was anticipated by the investigator
* Pregnant women Patients taking drugs that may slow down gastric Emptying such as: anticholinergic drugs, phenothiazines, antidepressants History of esophageal radiotherapy Unsubstituted hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Score for quality of visualization of the esophageal and gastric mucosa | During endoscopy
  The score is graded from A (good quality) to C (poor quality) according to a score developed by Elvas et al. (Endoscopy 2017).

SECONDARY OUTCOMES:
Questionnaire concerning security | During endoscopy
  Questionnaire filled by the investigator concerning the side effectets observed or not observed
Questionnaire concerning patient confort during fasting | The day of the endoscopy
  Snsations felt or not felt by the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No